CLINICAL TRIAL: NCT03444844
Title: Biodistribution and Dosimetry of Ga-68 P16-093 in Prostate Cancer Patients With Intermediate/High Risk Primary Disease or Biochemical Recurrence After Treatment
Brief Title: Biodistribution and Dosimetry of Ga-68 P16-093 in Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Five Eleven Pharma, Inc. (Industry)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IU-1711061247
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer Recurrent; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 68 Ga-P16-093

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Biochemical recurrent prostate cancer (Experimental): IV injection of 2 - 6 mCi of Ga-68 P16-093 followed by whole body PET/CT scanning (pelvis to shoulders) for ~ 60 min (~150 min for first 10 patients/dosimetry) starting immediately after injection.
  A contrast CT scan follows PET scan.
  Interventions: Drug: Ga-68 P16-093 PET/CT scan
- Intermediate/High Risk primary prostate cancer (Experimental): IV injection of 2 - 6 mCi of Ga-68 P16-093 followed by list mode PET/CT scanning using a fixed FOV including the pelvis area for ~ 50 min.
  Interventions: Drug: Ga-68 P16-093 PET/CT scan

INTERVENTIONS:
Drug: Ga-68 P16-093 PET/CT scan — IV injection followed by PET/CT scanning
  Other Names: PSMA-93; HBED-CC-PHENOXY-PSMA; PSMA-093; Ga-68-P16-093

SUMMARY:
Initial performance of Ga-68-P16-093 in prostate cancer patients including dosimetry and preliminary efficacy evaluation in BCR patients, and correlation of Ga-68-P16-093 uptake with tissue histopathology in intermediate to high risk primary prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria (Cohort 1):

* Male ≥ 18 years of age
* Prostate cancer patients presenting with rising PSA after radical prostatectomy for treatment if primary disease.
* PSA ≥ 0.2 ng/mL
* Patients must give informed consent for the research study, and agree to allow investigator access to clinical results following treatment plan implementation such as description of the treatment plan and PSA values following implementation of treatment plan as part of standard care, typically determined 3-4 months after treatment.

Inclusion Criteria (Cohort 2):

* Male ≥ 18 years of age
* Histologically confirmed prostate cancer with following Gleason scoring at biopsy:

  * Gleason ≥ 4+3 OR
  * Gleason 3+4 with >30% pattern 4 or ≥3 cores positive
* Scheduled for radical prostatectomy (expected to occur within 60-days of scanning)
* Patients must give informed consent for the research study, and agree to allow investigator access to the clinical results such as SOC imaging (mpMRI, e.g.) for surgical planning if done, or biopsy data following prostatectomy including lymph node dissection biopsy data, if available.

Exclusion Criteria (Cohorts 1& 2):

* Inability to give informed consent.
* Patient is unable to tolerate remaining still on the bed of the PET camera, due to physical limitations or claustrophobia.
* Significant acute or chronic medical, neurologic, or illness in the subject that, in the judgment of the Clinical Investigators, could compromise subject safety, limit the ability to complete the study, and/or compromise the objectives of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Ga-68-P16-093 in BCR | 2 weeks
  We will compare the number and location of metastatic lesions apparently detected by 68Ga-P16-093 with the number and location of lesions detected by standard-of-care imaging. Sensitivity of the 68Ga-P16-093 PET procedure will be estimated based on the number of subjects in whom a site of disease is identified by the imaging procedure. Scans will also be reconstructed summing passes 1-5, passes 2-5, passes 3-5, and passes 1-2 to assess how image quality varies with chosen framing.
The proportion of patients for whom Ga-18-P16-093 PET/CT changes treatment through detection of lesions | 4 months
  Change in management will be based on physician questionnaires including confirmation of actual treatment.
Sensitivity and Specificity of Ga-68-P16-093 in primary PCa | 2-60 days following PET/CT scan
  We will estimate the sensitivity and specificity of the 68Ga-P16-093 PET imaging by comparing the PET SUV values and whole-mount pathology findings on a sextant basis (6 sextants per subject x 10 subjects). Images will be evaluated from ~ 5 min to 60 minutes of scanning in 5-10 minutes up to 45 min frames.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Green, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Goodman Hall, Indiana Institute for Biomedical Imaging Sciences, Indiana University School of Medicine, Indianapolis, Indiana, United States